CLINICAL TRIAL: NCT05241327
Title: Effects of Nitrate-rich Beetroot Juice in Pregnant Women With High Blood Pressure
Acronym: NITBEETPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other); Novo Nordisk A/S (Industry); Danderyd Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Carlström, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DNR-2020-01596
Record Dates: First submitted 2022-02-05; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Preeclampsia; Hypertension; Endothelial Dysfunction; Nitric Oxide; Oxidative Stress; Proteinuria; Kidney Diseases
Keywords: Hypertension; Preeclampsia; Inorganic Nitrate; Endothelial dysfunction; Beetroot Juice
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Proteinuria; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial (RCT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Beetroot Juice (Nitrate, 400 mg)
  Interventions: Dietary Supplement: Beetroot Juice
- Placebo (Placebo Comparator): Beetroot Juice (Nitrate, 0 mg)
  Interventions: Dietary Supplement: Beetroot Juice

INTERVENTIONS:
Dietary Supplement: Beetroot Juice — Inorganic Nitrate
  Other Names: Beet It

SUMMARY:
BACKGROUND: Preeclampsia (PE) is a serious syndrome that affects 3-7% of all pregnant women. PE is characterized by hypertension and kidney problems after the 20th week of pregnancy and is associated with an increased risk of serious cardiovascular complications including death in both mother and fetus. The underlying disease mechanisms are not clear, but that there are changes in the vessels and their function is generally accepted. Today, there is a lack of medical treatment in the form of medicines.

HYPOTHESIS: So-called oxidative stress and deficiency of the vasodilator nitric oxide (NO) play an important role in disease onset and complications in PE.

WORK PLAN: This interdisciplinary project combines clinical and experimental studies to investigate the significance of oxidative stress and NO deficiency in PE. We have shown in previous studies that nitrate, which is found in high levels in lettuce and beets, can be converted to NO in the body. In a feasibility study, blood samples were taken from women with PE and healthy pregnant women. Analysis of these samples has shown that women with PE and their newborns have lower levels of nitrate and markers of NO in the blood. In a clinical study, the physiological effects (cardiovascular function, renal function, metabolic function) of an increased daily nitrate intake (in the form of a specially developed beetroot juice) are examined in patients with PE. Blood and urine samples are collected before and after beetroot intervention and during childbirth when umbilical cord and placenta samples are also collected. The samples are analyzed with biochemical analyzes with regard to e.g. oxidative stress and NO.

IMPORTANCE: The project is expected to contribute new and important knowledge regarding the disease mechanisms, which may enable new treatment strategies in PE.

DETAILED DESCRIPTION:
OVERALL PURPOSE:

1. Study the underlying disease mechanisms in preeclampsia Investigate the physiological effects of dietary nitrate in preeclampsia, in order to increase the production of nitric oxide in the body.

SPECIFIC GOALS:

Can increased intake of nitrate via the diet:

* increase the availability and function of nitric oxide?
* improve vascular function?
* lower blood pressure?
* reduce the morbidity of these patients and their newborns?

BACKGROUND:

Preeclampsia (PE) is a multi-system disorder characterized by hypertension, proteinuria and intrauterine growth restriction, affecting as many as 10% of healthy nulliparous women and is a major cause of morbidity and mortality in mothers, fetuses and newborns worldwide [1]. Cardiovascular disease and adverse complications (eg stroke and heart failure) are major causes of morbidity and mortality in pregnant women with PE. There are currently no approved treatment options available for PE patients, other than premature delivery. New studies on disease mechanisms are needed to improve the current treatment strategy in these high-risk patients.

The pathophysiology is complex and includes endothelial dysfunction, hypertension, renal failure, dyslipidemia and hypercoagulability. Several pathogenic mechanisms of PE have been postulated, but this remains to be fully elucidated. It is thought to be largely a result of dysfunction of the placenta, leading to increased uterine circulation resistance and uteroplacental hypoperfusion. This creates an ischemic / hypoxic placental environment that induces placental release of several pro-inflammatory and anti-angiogenic factors in the systemic circulation. These factors induce a systemic imbalance of redox status, altered angiogenic signaling, and a systemic inflammatory response, all of which induce and enhance extensive systemic endothelial dysfunction [2, 3]. It is this "second stage" of PE pathogenic consequences that is thought to contribute to its initial clinical findings. A key theory regarding the development and progression of PE-associated vascular endothelial dysfunction is increased production of angiotensin II and the formation of reactive oxygen species (ROS) as well as decreased efficiency of endogenous antioxidant systems, leading to a pro-oxidant state called oxidative stress. In addition, excessive ROS production limits the formation and bioactivity of nitric oxide (NO) from the enzyme NO synthase (NOS). NO is a vital molecule for the regulation of cardiovascular homeostasis via its modulation of vascular tone, platelet aggregation and renal function [4, 5]. During normal pregnancy, the NOS system is upregulated to promote a reduction in total peripheral resistance and blood pressure to allow adequate uteroplacental perfusion and fetal blood supply. Recent findings indicate that excessive ROS generation along with decreased NO signaling contribute to the pathogenesis of PE and associated cardiovascular complications [6]. New strategies that reduce oxidative stress and restore NO bioavailability during PE may therefore have therapeutic potential.

In addition to the L-arginine-dependent endothelial NOS (eNOS) pathway, there is another mechanism for NO generation, in which inorganic nitrate is serially reduced to form nitrite, NO and other bioactive NO-compounds in blood/tissues [7, 8]. Previously, nitrate was thought to be an inert circulating molecule in the blood that only reflected the degree of NO metabolism in the body. Accumulated evidence, however, shows that our daily diet is as important a source as NOS that contributes to the body's pool of this bioactive anion. Nitrate is found in high concentrations in vegetables, and especially in green-leafed lettuce, celery and beets. This type of food group has been associated with reduced cardiovascular risk in several clinical studies [9]. Previous findings have shown that dietary nitrate lowers blood pressure in healthy individuals [10] and hypertensive patients [11, 12]. Experimental studies show that nitrate can improve metabolic and kidney functions via mechanisms that include reduction of oxidative stress and restoration of NO [13]. The potential clinical significance of nitrate supplementation is of interest as the amounts of nitrate required for favorable cardiovascular effects may be obtained through our daily diet.

PROJECT DESCRIPTION:

* Population: Pregnant women will be included in the study from week 20 of pregnancy. Both pregnant women with blood pressure disease (such as PE, high blood pressure only during pregnancy and chronic high blood pressure) and healthy pregnant women with normal blood pressure will be examined.
* Design: Randomized, double-blind, placebo-controlled study with "on-treatment analysis of clinical trial data".
* Intervention: Study participants will be randomized to drink a beet juice (BEET-it-juice 70ml) that contains 400 mg of inorganic nitrate (Active juice) or beet juice without nitrate (Placebo juice) per day, for a total of 8-10 days. Study participants will receive the usual treatment and follow-up at the regular care unit. During the intervention period, patients are advised not to change their usual lifestyle (physical activity or diet). However, both groups should avoid nitrate-containing vegetables.
* Methods: A total of four research visits (about 2 hours each). Measurements and sampling will be made both before and after juice intake, and include blood pressure (office followed by 24 hours of continuous measurements), vascular function (flow-mediated dilation; FMD and microcirculation function, see descriptions below). Biological samples include blood and urine, which will be analyzed at Kliniskt Kem-Lab and used by our Laboratory at Biomedicum, KI Solna for various biochemical analyzes and functional studies.
* Blood pressure: Office blood pressure is measured in a sitting position (after 20 min of rest). Digital (automated) oscillometric apparatus is used and measurements are performed according to standardized protocol according to current guidelines. Outpatient blood pressure measurement (24 hours ABPM) is started after the end of the office measurement and is performed with a validated device (Model 90207, Spacelabs) Healthcare Ltd, Hertfordshire, UK) the day before and at the end of the juice intake period. During the day (07.00 - 23.00) a reading is made every 30 minutes and during the night (23.00 - 07.00) a reading is made every hour.
* FMD: A pen-like sensor is placed on the skin over a carotid artery just above the armpit, and the size of the blood vessel is measured for a few minutes. Then we inflate a small blood pressure cuff around the forearm for 4.5 minutes, and we measure again just when we release the pressure in the cuff. When the cuff is inflated, the patient may experience numbness of the hand, but this stops as soon as the air is released from the cuff. The procedure is completely harmless, and accepted method for evaluating endothelial function.

Microcirculation: Non-invasive, painless method where acetylcholine or nitroprusside are applied in a small chamber on the outside of the skin, and changes in the microcirculation are measured with laser speckle contrast analysis (LASCA) and with video microscopy at the nail fold. The method is painless and harmless. Uncommon but possible side effect is local rapid transient irritation of the skin.

The study participant will fill in a medicine journal to document ongoing blood pressure treatment during the study period, document the intake of the juice and fill in risk factors for developing blood pressure disease. Afterwards, a journal review of the birth outcome will be done to compare the maternal and fetal morbidity and mortality in both groups.

Population & Power: Primary clinical endpoints are lowering of systolic and diastolic blood pressure (office). Secondary endpoints are lowered blood pressure (24 hours ABPM) and improved endothelial function. Power calculation has been based on previous clinical studies in adult patients with hypertension and similar nitrate supplementation. Analysis based on 6% difference in blood pressure lowering between the groups, power (1-ß) of 0.80, type 1 error (α error rate) of 0.05, and standard deviation (σ) of 10% gave us a group size of at least n = 25 patients per group.

SIGNIFICANCE:

If the "NITBEETPE" study can show that morbidity is reduced through increased intake of dietary nitrate, it can enable new nutritional and future pharmacological treatment methods for PE. In the long run, it is hoped to find a safe and effective way to prevent the development of PE, which would of course be of great importance to many pregnant women and their children.

REFERENCES

1. B. Sibai, G. Dekker, M. Kupferminc, Pre-eclampsia, Lancet 365(9461) (2005) 785-99.
2. T. Chaiworapongsa, P. Chaemsaithong, L. Yeo, R. Romero, Pre-eclampsia part 1: current understanding of its pathophysiology, Nat Rev Nephrol 10(8) (2014) 466-80.
3. J.M. Roberts, C.A. Hubel, Is oxidative stress the link in the two-stage model of pre-eclampsia?, Lancet 354(9181) (1999) 788-9.
4. M. Carlstrom, C.S. Wilcox, W.J. Arendshorst, Renal autoregulation in health and disease, Physiol Rev 95(2) (2015) 405-511.
5. J.O. Lundberg, M.T. Gladwin, E. Weitzberg, Strategies to increase nitric oxide signalling in cardiovascular disease, Nat Rev Drug Discov 14(9) (2015) 623-41.
6. G. Osol, N.L. Ko, M. Mandala, Altered Endothelial Nitric Oxide Signaling as a Paradigm for Maternal Vascular Maladaptation in Preeclampsia, Curr Hypertens Rep 19(10) (2017) 82.
7. J.O. Lundberg, M. Carlstrom, F.J. Larsen, E. Weitzberg, Roles of dietary inorganic nitrate in cardiovascular health and disease, Cardiovasc Res 89(3) (2011) 525-32.
8. J.O. Lundberg, M.T. Gladwin, A. Ahluwalia, N. Benjamin, N.S. Bryan, A. Butler, P. Cabrales, A. Fago, M. Feelisch, P.C. Ford, B.A. Freeman, M. Frenneaux, J. Friedman, M. Kelm, C.G. Kevil, D.B. Kim-Shapiro, A.V. Kozlov, J.R. Lancaster, Jr., D.J. Lefer, K. McColl, K. McCurry, R.P. Patel, J. Petersson, T. Rassaf, V.P. Reutov, G.B. Richter-Addo, A. Schechter, S. Shiva, K. Tsuchiya, E.E. van Faassen, A.J. Webb, B.S. Zuckerbraun, J.L. Zweier, E. Weitzberg, Nitrate and nitrite in biology, nutrition and therapeutics, Nat Chem Biol 5(12) (2009) 865-9.
9. X. Wang, Y. Ouyang, J. Liu, M. Zhu, G. Zhao, W. Bao, F.B. Hu, Fruit and vegetable consumption and mortality from all causes, cardiovascular disease, and cancer: systematic review and dose-response meta-analysis of prospective cohort studies, BMJ 349 (2014) g4490.
10. F.J. Larsen, B. Ekblom, K. Sahlin, J.O. Lundberg, E. Weitzberg, Effects of dietary nitrate on blood pressure in healthy volunteers, N Engl J Med 355(26) (2006) 2792-3.
11. V. Kapil, R.S. Khambata, A. Robertson, M.J. Caulfield, A. Ahluwalia, Dietary nitrate provides sustained blood pressure lowering in hypertensive patients: a randomized, phase 2, double-blind, placebo-controlled study, Hypertension 65(2) (2015) 320-7.
12. V. Kapil, A.B. Milsom, M. Okorie, S. Maleki-Toyserkani, F. Akram, F. Rehman, S. Arghandawi, V. Pearl, N. Benjamin, S. Loukogeorgakis, R. Macallister, A.J. Hobbs, A.J. Webb, A. Ahluwalia, Inorganic nitrate supplementation lowers blood pressure in humans: role for nitrite-derived NO, Hypertension 56(2) (2010) 274-81.
13. M. Carlstrom, M.F. Montenegro, Therapeutic value of stimulating the nitrate-nitrite-nitric oxide pathway to attenuate oxidative stress and restore nitric oxide bioavailability in cardiorenal disease, Journal of internal medicine 285(1) (2019) 2-18.

ELIGIBILITY:
Inclusion Criteria:

Adult and decision-making patient who:

* is pregnant from week 20
* has normal blood pressure (controls) or high blood pressure during the current pregnancy (either chronic hypertension, gestational hypertension or preeclampsia)
* are cared for at Danderyd Hospital (Women's Clinic; Obstetrics and Gynecology)

Exclusion Criteria:

* Type 1 diabetes
* Vegetarians and vegans
* Regular use/need for proton pump inhibitors (PPi)
* Smoker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure (Office, Systolic) | 8-10 days supplementation with inorganic nitrate
  Reduction of office systolic pressure with 6%
Blood pressure (Office, Diastolic) | 8-10 days supplementation with inorganic nitrate
  Reduction of office diastolic pressure with 6%

SECONDARY OUTCOMES:
Blood Pressure (Mean Arterial Pressure, 24h ABPM) | 8-10 days supplementation with inorganic nitrate
  Reduction of Ambulatory Blood Pressure Monitoring (24 hours) with 6%
Endothelial function (Flow-mediated dilatation; FMD) | 8-10 days supplementation with inorganic nitrate
  Improved FMD response: Absolute increase of 1.1% (24% improvement from baseline)
Microvascular endothelium function (Laser Speckle Contrast Analysis; LASCA) | 8-10 days supplementation with inorganic nitrate
  Resistive Index (RI): absolute decrease in RI by 0.05 & relative decrease with 10%

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Carlstrom, PharmD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Karolinska_Institutet_Mattias_Carlstrom — https://staff.ki.se/people/mattias-carlstrom
- See also: Karolinska_Institutet_Josefine_Nasiell — https://staff.ki.se/people/josefine-nasiell
- See also: Karolinska_Institutet_Jonas_Spaak — https://staff.ki.se/people/jonas-spaak
- See also: Research_Gate_Josefine_Nasiell — https://www.researchgate.net/profile/Josefine-Nasiell-2
- See also: Research_Gate_Jonas_Spaak — https://staff.ki.se/people/jonas-spaak